CLINICAL TRIAL: NCT00513968
Title: A Single Center, Randomized, Open-label, Dose Escalating Phase I Study to Evaluate the Safety of Intramuscularly Administered DNA Vaccine (HB-110) Combined With Oral Antiviral (Adefovir) in Subjects With Chronic Hepatitis B Over a 48-week Period
Brief Title: Phase I Study to Investigate the Safety and Efficacy of HBV DNA Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB110_HB_I
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): HB-110 2mg, 4mg or 8mg combined with Adefovir
  Interventions: Genetic: a mixed plasmid DNA (HB-110)
- II (Active Comparator): Adefovir
  Interventions: Drug: Adefovir

INTERVENTIONS:
Genetic: a mixed plasmid DNA (HB-110) — HB-110 2mg (or 4mg or 8mg), im, every other week, from week 0 to week 22 (total 12 injections) and Adefovir(Adefovir dipivoxil 10mg), od, from week -10 to from week 48.
  Arms: I
Drug: Adefovir — Adefovir(Adefovir dipivoxil)10mg, od, from week -10 to week 48.
  Arms: II

SUMMARY:
This study will evaluate the safety and immunogenicity of a novel mixed plasmid DNA (HB-110) combined with an antiviral agent (Adefovir) for the patients with chronic Hepatitis B infection.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B infected patient documented with positive HBsAg for 3 months and more at screening
* Chronic hepatitis B infected patient with positive HBeAg at screening
* Patient who has not treated with interferon alpha, lamivudine or adefovir within 3 months before study entry
* HBV DNA more than 1x10^5 copies/mL through COBAS Amplicor HBV monitor assay or bDNA method at screening
* Patient with HBV DNA decrease more than 10-fold compared to the baseline after 8 weeks treatment with adefovir
* Patient with ALT value between ULN x 1.5 and ULN x 5 at screening
* Patient given a written consent voluntarily

Exclusion Criteria:

* Have uncompensated liver disease
* Serum creatinine > ULN x 1.5
* Are positive for Hepatitis C, hepatitis D or HIV infection (confirmed by ELISA assay)
* Had a previous liver or bone marrow transplant
* Are currently taking any immunosuppressant or any possible immune modulatory drugs
* Women who are pregnant or breastfeeding
* Woman or man who plans a birth for study duration
* Any experience of severe adverse drug reaction or any medical history of severe allergic disease
* Patient with any severe disease (for example, heart failure, renal failure, pancreatitis, diabetes mellitus) affecting the study in discretion of investigator except liver disease
* Patient with any other liver disease but hepatitis B (for example, hemochromatosis, Wilson's disease, alcoholic/non-alcoholic liver diseae)
* Patient with intrahepatic tumors confirmed by imaging (liver biopsy)and abnormally increased alpha-fetoprotein
* Patient with any present malignant tumor except liver or its history
* Other inappropriate patient in discretion of investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2007-07; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adverse events and clinical laboratory abnormalities | 48 weeks

SECONDARY OUTCOMES:
HBeAg/HBsAg seroconversion rate, HBV Ag specific T cell immunity | 24, 28, 32, 42, 44, and 48 week

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Seung-kyu Yoon, M.D., Principal Investigator — The Department of Gastroenterology at Seoul St. Mary's Hospital
Locations (1):
- Kangnam St. Mary's Hospital, Seoul, South Korea